CLINICAL TRIAL: NCT05268406
Title: Evaluation of C-Scan in Identifying Subjects With Elevated Risk of Polyps in the Colon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Check-Cap Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CL-SY-01-0099
Record Dates: First submitted 2022-02-15; First posted 2022-03-07 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-02

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): All study participants will undergo the C-Scan System procedure, followed by a standard of care optical colonoscopy
  Interventions: Device: C-Scan System

INTERVENTIONS:
Device: C-Scan System — Subjects will be provided with contrast agent and dietary fiber pills, and instructed to start intake approximately 48 hours prior to the planned C-Scan procedure start. C-Scan system intervention includes ingestion of the C-Scan Cap and attachment of the C-Scan track to the subject's lower back. The subject is required to keep the C-Scan Track attached to the lower back and to continue intake of contrast agent and dietary fiber pills until the C-Scan Cap's natural excretion. Standard of care optical colonoscopy will be performed within 60 days from the C-Scan Cap ingestion.

SUMMARY:
The purpose of the first part of the study (subgroup R&D) is to demonstrate the safety and performance of the C-Scan system and to collect data in order to improve the analysis process. The purpose of the second part of the study (subgroup pre-pivotal) is to determine the ability of the C-Scan System to identify elevated risk subjects

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female at the age of 50-75 years old
2. Able to provide a signed informed consent.
3. Willing and able to comply with the specified study requirements and can be contacted by telephone.
4. Scheduled for colonoscopy procedure within 60 days of C-Scan ingestion within the research institution's system.*
5. Maximum body (abdominal) circumference < 125 cm.

Exclusion Criteria:

1. Subject who is not a suitable candidate for a colonoscopy
2. Known history of dysphagia or other swallowing disorders.

   Third (3rd) and fourth (4th) exclusion criteria are applicable to the pre-pivotal subgroup only:
3. History of the following:

   * Previous colon polyps
   * Personal history of CRC
   * Family history of CRC or adenomatous polyps diagnosed in a relative before age 60 years
   * History of inflammatory bowel disease
   * Having an inherited syndrome (Lynch syndrome, FAB)
4. GI bleeding within the last 3 months i.e., rectal outlet bleeding, hematochezia or melena
5. Known motility disorders:

   1. Chronic Constipation: less than three (3) bowel movements/week, without the use of laxatives within the last 3 months.
   2. Delayed gastric emptying.
   3. Ongoing diarrhea defined as passage of loose or watery stools at least three times in a 24-hour.
6. Known IBD (Crohn's, ulcerative Colitis)
7. Prior history of gastrointestinal tract surgery.
8. Prior history of abdominal surgery that might cause bowel strictures leading to capsule retention, as determined by physician discretion.
9. Any condition believed to have an increased risk for capsule retention, known strictures, any prior episode of bowel obstruction: known bowel adhesion, any 'obstacles' to free passage of the capsule (such as intestinal tumors, radiation enteritis) or incomplete colonoscopies or incomplete colonoscopies as determined by physician discretion.
10. Significant change in diameter and frequency of stool within the last 3 months
11. Has an implanted cardiac device or any other implanted active device
12. Known sensitivity to iodine or hyperthyroidism
13. Acute kidney failure
14. Known condition which precludes compliance or is contraindicated with study and/or device instructions.
15. Has any procedure requiring contrast agent or which may introduce electronic interference (such as magnetic resonance imaging, DEXA scan) or an imaging procedure pre-scheduled within 14 days of C-Scan ingestion
16. Nuclear imaging procedure during 4 weeks before C-Scan procedure
17. Known condition of opioid use disorder and/or alcoholism.
18. Women who are either pregnant or nursing at the time of screening (to be verified by urine or serum pregnancy test for woman of child- bearing potential who are not post-menopausal or undergone surgical sterilization(
19. Concurrent participation in another clinical trial using any investigational drug or device.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Determine the ability of the C-Scan System to identify elevated risk subjects | 60 days
  Sensitivity for detecting subjects with elevated risk for polyps
Determine the ability of the C-Scan System to identify elevated risk subjects | 60 days
  Specificity for detecting subjects with elevated risk for polyps

SECONDARY OUTCOMES:
Incidence of device or procedure related adverse events | Up to 7 days post C-Scan procedure completion
  Analysis of safety data
Satisfaction with the C-Scan procedure assessed by a questionnaire | Up to 7 days post C-Scan procedure completion
  Satisfaction questionnaire to be completed by the subject
Satisfaction with the C-Scan procedure compared to colonoscopy assessed by a questionnaire | Up to 7 days post colonoscopy
  Satisfaction questionnaire to be completed by the subject
Evaluate the Whole Gut Transit Time | During the C-Scan procedure
  Time elapsed from capsule ingestion to excretion

CONTACTS AND LOCATIONS:
Overall Officials: Nadir Arber, Professor, Principal Investigator — Tel Aviv Medical Center, Israel
Locations (10):
- Israel (10):
  - Emek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Bnei Zion Medical center, Haifa
  - Lin- Clalit, Haifa
  - Rambam Medical Center, Haifa
  - Talpiot- Clalit, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galil Medical Center, Nahariya
  - Laniado Medical Center, Netanya
  - Tel Aviv Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No